CLINICAL TRIAL: NCT06632548
Title: Retention of Three Different Secondary Copings in Telescopic Attchments Used to Stabilize Implant Retained Mandibular Overdenture a Randomized Clinical Trial
Brief Title: Retention of Three Different Types of Telescopic Attachments
Acronym: Overdenture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Moatz Aly Ahmed Hussien (Other)
Responsible Party: Sponsor-Investigator, Moatz Aly Ahmed Hussien, Assistant lecturer at prosthodontic department, Beni-Suef University
Organization: Beni-Suef University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 612
Record Dates: First submitted 2024-10-07; First posted 2024-10-09 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2022-07

CONDITIONS: Edentulism; Denture Retention
Keywords: overdenture-telescopic attachment-poly ether ketoneketone-PEKK-; milled titanium; 3d printed cobalt chromium; implant retained overdenture; mandibular overdenture

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- milled titanium secondary coping (Active Comparator): group I patients received primary and secondary coping made of milled titanium
  Interventions: Device: telescopic overdenture
- 3D printed cobalt chromium secondary coping (Experimental): group II patients received primary coping made of milled titanium and secondary coping made of 3D printed cobalt chromium
  Interventions: Device: telescopic overdenture
- milled poly ether ketone ketone secondary coping (Experimental): group III patients received primary coping made of milled titanium and secondary coping made of milled poly ether ether ketone
  Interventions: Device: telescopic overdenture

INTERVENTIONS:
Device: telescopic overdenture — two implant retained mandibular overdenture with telescopic attachment

SUMMARY:
This study was conducted on thirty patients. These patients were divided into three groups in a random manner to compare the retention forces between three different types of secondary crowns used to stabilize two implant mandibular overdentures. in all groups the primary coping was fabricated from milled titanium while the secondary coping was milled titanium in first group ,3D printed cobalt chromium in the second group and milled poly ether ketone ketone in the third group the retention forces was measured using forcemeter immediately after insertion and after 3,6, months

DETAILED DESCRIPTION:
A thirty edentulous patients Was selected from outpatient clinic of

Exclusion criteria:

1. systemic and metabolic disorders that may complicate osseointegration.
2. Patients receiving bisphosphonates.
3. patients receiving radiotherapy. The patients was assigned into three groups using balanced randomly. Patients was randomly allocated into one of three groups using random numbers generated using Excel program.

Group I included patients who received 2 implants and telescopic overdentures with milled titanium primary and secondary coping Group II included patients who received telescopic overdentures with milled titanium primary coping and three dimensionally printed secondary coping GroupIII patients recived milled titanium primary coping and poly ether ketone ketone secondary copings (PEKK) secondary coping All patients signed an informed consent.

Surgical and prosthetic protocols:

A radiographic stent with gutta percha markers at the canine region was fabricated and the patient was instructed to wear it during cone beam radiographic evaluation to evaluate proposed implant sites regarding bone height and thickness, and approximation to vital structures (mental foramen).

Radiographic template was converted to surgical template.

The two implants was inserted nearly parallel as possible. If inclination of the implants was inevitable buccally or lingually due to mandibular concavities, the inclination was compensated later during design of primary copings.

The implants was inserted in the canine region with two steps surgical protocol. After three months of the insertion and osseointegration implants was exposed and healing abutments was inserted after gingival healing implant level impression will be taken.

The metallic primary coping was milled with 2-degree convergence for all cases while the second coping was milled titanium or 3D printed cobalt chromium or milled PEKK according the patient group.

the primary copings was screwed to the implants and the secondary coping pick up was done and patient was instructed to follow oral hygiene measures and was scheduled for periodic follow up every 3 months.

Evaluation of overdenture retention:

Force meter device was used to measure the retention of the mandibular overdenture in Newton.

The patient was seated on upright position and asked to open his mouth until the occlusal surface of the lower denture is parallel to the floor and the maximum dislodging force to remove the denture is recorded using digital forcemeter.

Measurement of retention forces was made immediately after overdenture insertion and repeated at 3,6,9and 12 months after insertion after by independent dental personnel blinded to treatment groups.

ELIGIBILITY:
Inclusion Criteria:

1. un-satisfaction with the retention of mandibular dentures due to mandibular ridge atrophy and desired to have more stable prosthesis,
2. sufficient remaining bone in height, width and thickness in the interforaminal area to allow installation of at least 3.5mm diameter implants.
3. Adequate amount of interarch space of at least 12mm from the occlusal plane of the mandibular denture to the mucosa of the ridge. Patients with the 4- age range 55 to 75 years.

   -

   Exclusion Criteria:

1) systemic and metabolic disorders that may complicate osseointegration. 2) Patients receiving bisphosphonates. 3) patients receiving radiotherapy.

-

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-08-30 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-03-30 (Actual)

PRIMARY OUTCOMES:
retention forces | from insertion time up to one year follow up
  retention forces of three different type secondary coping telescopic attachments used to stabilize two implant mandibular overdenture these attachments are made of either milled titanium, 3D printed cobalt chromium or milled poly ether ketone ketone

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry Minia University, Elminia, Elminia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
the values of retention of each individual plus age and sex
Supporting Information: Study Protocol, SAP, CSR
Time Frame: starting after release of the research publication and ending after one year
Access Criteria: any researcher interested in the prosthodontics can ask for IPD will be able to ask for the participant individual data relating to their results,age,sex and planning of the case
URL: https://dent.bsu.edu.eg/homepage.aspx?Pid=1844